CLINICAL TRIAL: NCT05763355
Title: Multicentric Comparative Prospective Study of the Benefits and Risks of Biopsy Prostate Using Transrectal or Transperineal Procedure for the Prostate Cancer Diagnostic.
Acronym: BIOPROSTABORD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-A02436-35
Record Dates: First submitted 2023-01-11; First posted 2023-03-10 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Patients With Suspected Prostate Cancer
Keywords: Transpérinéal; Transrectal; Biopsy; Prostate; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transrectal biopsy using KOELIS fusion system (Other): Transrectal procedure will be performed with the patient in the left lateral position with a completely free-hand technique utilising the KOELIS fusion system.
  Interventions: Procedure: Biopsy
- Transperineal biopsy using KOELIS perine grid (Other): Transperineal biopsy will be performed in the lithotomy position. KOELIS "Perine Grid" needle guidance device and "Steady Pro" free-hand probe arm will be utilised (free-hand assisted technique).
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — Biopsies will be performed under local anaesthesia. In all patients with a suspicious lesion (PIRADSv2.1 3-5) noted on the mp-MRI, the software-based image fusion biopsies will be obtained collecting 3 to 5 cores per target area according to its volume, 10-12 systematic cores of the remaining areas of the prostate will be collected from sectors specified in the PIRADSv2.1 prostate map.

SUMMARY:
The performance of prostatic biopsies is an essential element to confirm the diagnosis of prostate cancer and to specify the characteristics of the tumor in terms of stage and grade.

The first route of prostatic biopsies is mainly transrectal with passage of a needle introduced into the guide fixed on the endorectal ultrasound probe. There is another possible access route, transperineal, with prostatic puncture by a needle introduced transcutaneously, guided by an endorectal ultrasound image. The first transperineal route would offer the first benefit for the patient, to reduce the infectious risk inherent in the endorectal way. It would also reduce the risk of rectal bleeding.

In addition, the transperineal pathway appears to be able to improve the detection threshold of prostatic tumours located on the anterior part of the gland due to the angle of penetration of the needle and its more anterior positioning relative to the prostate.

There is currently no randomized comparison study of the transperineal versus transrectal procedure on infectious risk. The aim of the project is to enable this comparative study, within our institution where experienced urologist surgeons practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected prostate cancer with at least one of the following criteria met :

  1. MRI Staging: T2 or T3a,
  2. MRI Grading: Pirads greater than or equal to 3
  3. MRI tumor volume greater than or equal to 0.5 cm3

  e.Patient without tumor lesion detected by prostate MRI less than 3 months old with PSA > 4 ng/ml, or an observed suspicious induration to the rectal exam
* Voluntarily signed and dated written informed consents prior to any study specific procedure,

Exclusion Criteria:

* Other medical conditions may interfere with the conduct of the study and, in the judgment of the investigator, would make the patient inappropriate for entry into this study,
* Individuals deprived of liberty or placed under legal guardianship,
* Unwillingness or inability to comply with the study protocol for any reason.
* Patients without a health insurance

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 596 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of the rate of occurrence of biopsy-induced infection in both groups | 30 days after intervention
  Biopsy-induced infection are defined as :
  * Positive post-biopsy urinary test result
  * Clinical infection syndrome (T>37.5°C fever)
  * Signs of urogenital infection (cystitis/prostatitis/orchi-epididymitis)
  * Hospitalization for hyperpyrexia
  * Septic shock

SECONDARY OUTCOMES:
Comparison of the rate of rectal bleeding in both groups | 30 days after intervention
Comparison of the rate of urethral bleeding (hematuria and urethrorrhagia) in both groups | 30 days after intervention
Comparison of the percentage of negative biopsies in both groups | 30 days after intervention
Comparison of the percentage of positive biopsies on on anterior areas in both groups | 30 days after intervention
Comparison of the Percentage of underestimation of the stage of tumor development in both groups | 3 months after intervention
  Confrontation with the MRI result and the resected specimen of the radical prostatectomy
Assess the pain (tolerance) felt by the patient according to the biopsy method used | 1 day
  EVA pain scale at J0
Comparison of the Room occupancy time in both groups | 1 day
Comparison of the Procedure Time in both groups | 1 day
  Procedure time = Endorectal Ultrasound Probe Introduction Time - Probe Removal Time
Comparison of the Average Length of Stay in both groups | 1 day

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Clinique St Augustin, Bordeaux
  - Centre Médico-Chirurgical Les Cèdres, Brive-la-Gaillarde